CLINICAL TRIAL: NCT02926027
Title: Effect of Vascepa on Progression of Coronary Atherosclerosis in Persons With Elevated Triglycerides (200-499) on Statin Therapy
Brief Title: Effect of Vascepa on Improving Coronary Atherosclerosis in People With High Triglycerides Taking Statin Therapy
Acronym: EVAPORATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Intermountain Research and Medical Foundation (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21733-01
Record Dates: First submitted 2016-09-28; First posted 2016-10-06 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active subjects (Active Comparator): Vascepa (4 gm/day), oral dose
  Interventions: Drug: Vascepa
- Placebo subject (Placebo Comparator): oral dose of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vascepa — Vascepa is a an Eicosapentaenoic acid (EPA), an omega-3 polyunsaturated fatty acid.
  Other Names: icosapent ethyl
  Arms: Active subjects
Drug: placebo — placebo
  Arms: Placebo subject

SUMMARY:
Effect of Vascepa on Progression of Coronary Atherosclerosis in Persons with Elevated Triglycerides (200-499) on Statin Therapy. The study is to determine progression rates of low attenuation plaque under influence of Vascepa as compared to placebo.

DETAILED DESCRIPTION:
Residual cardiovascular (CV) risk remains in dyslipidemic patients despite intensive statin therapy, underscoring the need for additional intervention. Eicosapentaenoic acid (EPA), an omega-3 polyunsaturated fatty acid, is incorporated into membrane phospholipids and atherosclerotic plaques and exerts beneficial effects on the pathophysiologic cascade from onset of plaque formation through rupture. EPA also improves atherogenic dyslipidemia characterized by reduction of triglycerides without raising low-density lipoprotein cholesterol. All of this data supports the biologic plausibility of EPA as an anti-atherosclerotic agent. The goal of this study is to evaluate whether treatment with Vascepa (4 grams) results in a greater change from baseline in low attenuation plaque than placebo in subjects with elevated triglycerides (200-499 mg/dl).

ELIGIBILITY:
Inclusion Criteria:

* Elevated triglycerides (fasting value between 200-499 mg/dl) at qualifying or baseline visit.
* LDL-C ≤115 mg/dL on appropriate statin therapy
* LDL-C >40 mg/dL
* Stable diet and exercise, as defined as the same pattern for the previous 4 weeks
* Stable treatment with a statin+/- ezetimibe for at least 4 weeks
* Patients with at least 1 angiographic stenosis with at least 20% narrowing by coronary computed tomography angiography (CTA).
* Willingness to be on birth control for women of childbearing age or established post-menopausal

Exclusion Criteria:

* A contraindication to fish or fish oils including: known hypersensitivity to drug or fish.
* Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator or principal investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study.
* Non-study lipid altering medications or supplements (ie - Niacin, PCSK9, fibrates, bile acid Sequestrants, dietary fish oil supplement capsules, orlistat [OTC (Alli®) as well as Rx (Xenical®)] or other drugs used for weight loss).
* Stable (same daily dose for the last 4 weeks) on medications that can affect lipids (retinoids, hormones, steroids, HIV medications, chemotherapy, thyroid medications).
* BMI > 40
* Bleeding disorder
* Uncontrolled hypertension (SBP≥ 180 mmHg or DBP≥100 mmHg)
* History of known myocardial infarction, stroke or life-threatening arrhythmia within the prior six months.
* NYHA Class III- IV heart failure
* History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy.
* Serum creatinine > 1.4 mg/dl
* Drug or alcohol abuse, or current intake of more than 14 ounces of alcohol per week for men and 10 ounces for women
* Concurrent enrollment in another placebo-controlled trial or within 30 days of finishing another trial
* Partial ileal bypass or known gastrointestinal disease limiting drug absorption
* History of hypertensive encephalopathy or cerebrovascular accident
* Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator or PI
* Pregnancy
* Genetic mutations/polymorphisms having an effect on blood lipids
* History of coronary artery bypass surgery
* Allergy to contrast material
* Allergy to beta-blocker in subjects with resting heart rate >70 bpm

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation (The Lundquist Institute)
Locations (2):
- United States (2):
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center (The Lundquist Institute), Torrance, California
  - Intermountain Medical Center, Intermountain Heart Institute, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data will be tabulated and analysed. Study site will not share any of the subject identifiers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Subjects | Placebo Subject
Started | 40 | 40
Completed | 31 | 37
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Subjects | Placebo Subject | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 31 | 61
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.9) | 58.3 (8.6) | 57.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 22 | 45
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 33 | 33 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Progression Rates of Low Attenuation Plaque Under Influence of Vascepa as Compared to Placebo as a Change Between Two or More Time Points
Description: low attenuation plaque volume change from baseline to 18 months
Time Frame: 18 months
Population: completed study
Measure: Mean (Standard Deviation); unit: volume in mm cubed
Arm/Group | Active Subjects | Placebo Subject
Number analyzed (Participants) | 31 | 37
volume in mm cubed | -0.3 (1.5) | 0.9 (1.7)

2. Secondary Outcome: The Composition of Non-calcified Coronary Atherosclerotic Plaque (NCP)
Description: the measure is reported as volume of non-calcified plaque, as the secondary measure has been reported.
Time Frame: 18 months
Population: all participants finishing final CT angiogram
Measure: Mean (Standard Deviation); unit: MM CUBED
Arm/Group | Active Subjects | Placebo Subject
Number analyzed (Participants) | 31 | 37
MM CUBED | -0.8 (1.2) | 0.3 (1.3)

ADVERSE EVENTS:
Time Frame: 18 month follow up
Arm/Group | Active Subjects | Placebo Subject
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT02926027/Prot_SAP_001.pdf